CLINICAL TRIAL: NCT05870007
Title: Atorvastatin and Alkali Therapy in Patients With Autosomal Dominant Polycystic Kidney Disease, A Pilot Trial for Safety and Feasibility
Brief Title: Atorvastatin and Alkali Therapy in Patients With Autosomal Dominant Polycystic Kidney Disease
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: Taipei Medical University Shuang Ho Hospital (Other)
Collaborators: University of Southern California (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TMU-JIRB N202208049
Record Dates: First submitted 2023-04-12; First posted 2023-05-23 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2023-01

CONDITIONS: Autosomal Dominant Polycystic Kidney Disease; Chronic Kidney Diseases
MeSH Terms: conditions — Polycystic Kidney, Autosomal Dominant; Renal Insufficiency, Chronic | interventions — Atorvastatin; Tablets; Sodium Bicarbonate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control group (No Intervention): Standard treatment alone
- Atorvastatin (Active Comparator): Standard treatment + Atorvastatin 20mg QD
  Interventions: Drug: Atorvastatin 20 Mg Oral Tablet
- Atorvastatin AND Alkali (Active Comparator): Standard treatment + Atorvastatin 20mg QD + Sodium Bicarbonate therapy up to 1800mg per day
  Interventions: Drug: Atorvastatin 20 Mg Oral Tablet; Drug: Sodium Bicarbonate 600 Mg Oral Tablet

INTERVENTIONS:
Drug: Atorvastatin 20 Mg Oral Tablet — Atorvastatin 20mg
  Arms: Atorvastatin; Atorvastatin AND Alkali
Drug: Sodium Bicarbonate 600 Mg Oral Tablet — Sodium bicarbonate would be titrated up to 1800mg per day according to metabolic acidosis severity during clinical follow-up
  Arms: Atorvastatin AND Alkali

SUMMARY:
Polycystic Kidney Disease (PKD) is the most common genetic disease leading to End Stage Kidney Disease (ESKD), affecting between 1 in 500-1000 individuals from every ethnic group. The autosomal dominant (ADPKD) form arises from a two-hit downregulation of proteins encoded by either PKD1 or PKD2. Although many potential therapies have been studied to slow progression of ADPKD, none to date have been proven to be both safe and effective in slowing disease progression. Cholesterol-lowering agents called statins have shown promise in the treatment of younger ADPKD patients, reducing inflammation and progression as assessed by kidney growth, but their utility appears to be limited in older populations and those with more advanced chronic kidney disease (CKD). Recent evidence suggests that acidosis, as often seen in patients with worsening CKD and which may enhance CKD progression, limits the effectiveness of statins and enhances their potential toxicity. The investigators thus hypothesize that correction of acidosis along with statin treatment will be a safe and effective therapeutic regimen to slow CKD progression in the adult ADPKD population and improve overall quality of life in these patients. To test this hypothesis, the investigators will conduct a pilot open-label randomized clinical trial in ADPKD patients with estimated GFR >45 min (Stage 1-3a CKD) comparing three treatment groups: control, atorvastatin (20 mg po qd), and atorvastatin plus sodium bicarbonate tablets (upto 1800mg po total daily dose) over one year. At the beginning of the study, the investigators will determine the genotype of the trial participants. During the study period, through study visits along with serial blood draws and urinary measurements, the investigators will evaluate safety and tolerability of these treatment regimens, follow renal function and investigate the role of these treatments on acidosis, inflammatory and metabolic biomarkers in patients enrolled at an outpatient facility. Serial follow-up imaging study will also be done in selected patients. This study will establish the framework for larger clinical trials in ADPKD. Moreover, if the results of this study suggest safety/tolerability or potential benefits of statins and alkali therapy in this ADPKD population, the investigators will seek extramural funding for a larger clinical trial to test this therapeutic strategy in ADPKD.

ELIGIBILITY:
Inclusion Criteria:

1. Patient voluntarily gives informed consent to participate in the study and signed study's IC and HIPAA.
2. Patient is age 18 or older at the time of consent.
3. If applicable, female of reproductive potential (Females who are successfully sterilized (surgical sterilization methods include hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or are postmenopausal (defined as amenorrhea for at least 12 consecutive months) are not considered to be of reproductive potential) must be non-pregnant (as confirmed by a urine pregnancy test at screening) and non-lactating, and agree:

   1. Either abstain from intercourse (when it is in line with their preferred and usual lifestyle), or
   2. Use 2 medically acceptable, highly-effective forms of contraception for the duration of study, and at least 30 days after discontinuing study drug (highly-effective forms of contraception can include approved hormonal contraceptives (oral, injectable, and implantable), and barrier methods (such as a condom or diaphragm) when used with a spermicide.))
4. Patients has ADPKD diagnosed by unified criteria using a combination of ultrasound results, genotyping and MRI as needed (1, 2). Kidney ultrasound is usually used for screening because it is safe, effective, and inexpensive. Diagnostic criteria are based upon whether the genotype is known. Disease severity varies between the different genotypes. The great majority of patients at risk for ADPKD are from families with an unknown genotype. This diagnosis will take place prior to recruitment / inclusion into the study.

   The following ultrasonographic criteria for the diagnosis of ADPKD are for at-risk patients from families of where the genotype is not known:
   1. If the patient is between 18 and 39 years of age, at least three unilateral or bilateral kidney cysts. The specificity and positive predictive value at this age-range is 100 percent. (sensitivity of 82 and 96 percent for individuals between 15 and 29 years and between 30 to 39 years of age, respectively).
   2. If the patient is 40 to 59 years of age, at least two cysts in each kidney (sensitivity, specificity, and positive predictive value of 90, 100, and 100 percent, respectively).
   3. Among individuals 60 years or older, at least four cysts in each kidney. (100 percent sensitivity and specificity).
5. The above patients with estimated GFR ≥30 ml/min i.e. with stage 1-3b CKD
6. Plasma bicarbonate ≤ 25 mMol/L
7. Metabolic acidosis
8. The patient agrees to immediately inform Investigator and research coordinator of any changes or planned changes in concomitant medication

Exclusion Criteria:

1. Patients with known allergy or sensitive to Atorvastatin or NaHCO3
2. Acute coronary disease, liver disease, muscle disease, or a history of pulmonary edema
3. Creatine Phospho Kinase (CPK) > 2ULN (2.5 ULN in African Americans). Elevated creatine phosphokinase could be a marker of rhabdomyolysis, which is a potential side effect of pravastatin. In general, patients with African American ancestry can have higher normal level of CPK
4. Patients with systemic disease that impacting kidney per Investigator's decision
5. Patients with known unstable cerebral aneurysm per Investigator's decision
6. Pregnancy or lactation, or patients who refuse to use recommended contraception methods
7. Proteinuria > 1000 mg/day
8. History of non-compliance of medication per Investigator's decision
9. Patients with uncontrolled hypertension, edema, or development of severe MA as per Investigator's decision
10. History of cancer
11. History of liver disease: hepatic failure/shock, cirrhosis
12. Current or planned use of any of prohibited concomitant medication
13. Patients with history of nephrolithiasis

Following medications prohibited at the time of enrollment and during the study and if the patient is started on these medications then the patient will be excluded from the study:

rapamycin or its analogues tolvaptan spironolactone cimetidine and ketoconazole erythromycin cyclosporine gemfibrozil colchicine niacin (>1 g/day) other lipid lowering medications in the class of statins

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-05 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Changes in kidney function in patients enrolled in different arms of the study | 12 months
  The investigators will estimate the effect of Atorvastatin and NaHCO3 on kidney function in patients with ADPKD compared to Atorvastatin alone or Standard therapy: serum creatinine-derived estimated glomerular filtration rate (eGFR) calculated by CKD-EPI equation, to evaluate kidney function.
Changes in kidney function in patients enrolled in different arms of the study | 12 months
  The investigators will estimate the effect of Atorvastatin and NaHCO3 on kidney function in patients with ADPKD compared to Atorvastatin alone or Standard therapy: serum blood urea nitrogen (BUN), to evaluate kidney function.
Changes in kidney function in patients enrolled in different arms of the study | 12 months
  The investigators will estimate the effect of Atorvastatin and NaHCO3 on kidney function in patients with ADPKD compared to Atorvastatin alone or Standard therapy: serum sodium level (Na), to evaluate kidney function.
Changes in kidney function in patients enrolled in different arms of the study | 12 months
  The investigators will estimate the effect of Atorvastatin and NaHCO3 on kidney function in patients with ADPKD compared to Atorvastatin alone or Standard therapy: serum potassium level (K), to evaluate kidney function.
Changes in liver function in patients enrolled in different arms of the study | 12 months
  The investigators will test liver function test panels in patients with ADPKD compared to Atorvastatin alone or Standard therapy. The liver function panel should be within normal limits for enrollment and continuation in the study. Liver function test with ALT will be evaluated at the end of the trial.
Changes in liver function in patients enrolled in different arms of the study | 12 months
  The investigators will test liver function test panels in patients with ADPKD compared to Atorvastatin alone or Standard therapy. The liver function panel should be within normal limits for enrollment and continuation in the study. Liver function test with AST will be evaluated at the end of the trial.
Changes in liver function in patients enrolled in different arms of the study | 12 months
  The investigators will test liver function test panels in patients with ADPKD compared to Atorvastatin alone or Standard therapy. The liver function panel should be within normal limits for enrollment and continuation in the study. Liver function test with total bilirubin will be evaluated at the end of the trial.
Changes in liver function in patients enrolled in different arms of the study | 12 months
  The investigators will test liver function test panels in patients with ADPKD compared to Atorvastatin alone or Standard therapy. The liver function panel should be within normal limits for enrollment and continuation in the study. Liver function test with increase in prothrombin time will be evaluated at the end of the trial.
Changes in muscle injury marker function in patients enrolled in different arms of the study | 12 months
  The investigators will estimate the effect of Atorvastatin and NaHCO3 on creatine phospho kinase (CPK) in patients with ADPKD compared to Atorvastatin alone or Standard therapy.
Changes in muscle tenderness in patients enrolled in the study | 12 months
  The investigators will estimate the effect of Atorvastatin and NaHCO3 on muscle tenderness in patients with ADPKD compared to Atorvastatin alone or Standard therapy. The physical exam will evaluate tenderness to palpation in major muscle groups such as leg, arm and back muscles. It will be graded as presence or absence. The patients will only be enrolled if there is absence of tenderness in muscles upon palpation on physical exam. If there is tenderness on exam or the patient reports tenderness that is then confirmed by exam the patient will be removed from the study.
Changes in blood pressure in patients enrolled in different arms of the study | 12 months
  The investigators will estimate the effect of Atorvastatin and NaHCO3 on blood pressure (systolic and diastolic) in patients with ADPKD compared to Atorvastatin alone or Standard therapy

SECONDARY OUTCOMES:
Urinary alkalinization changes | 12 months
  These parameters will be ascertained by measurements of urinary pH.
Inflammatory markers in blood and urine | 12 months
  The investigators will assess inflammatory markers (interleukins, prostaglandins and other cytokines) in leukocytes, plasma, and urine in the different study groups.
  The biomarkers that will be measured are
  HETE / HODE species phospho-AMPK Inflammatory and metabolic biomarkers: NGAL, KIM1 in blood and urine.
AMPK pathway activation | 12 months
  The investigators will determine whether and to what extent the AMPK pathway is activated in leukocytes and urine derived from patients in the study groups at the different study visits. Concentration of AMPK pathway-related metabolites in serum and urine would be measured (Creatinine, Osmolality, Lactate, Pyruvate, Succinate, Total Protein, PKM2, LDHA, PDK1).

CONTACTS AND LOCATIONS:
Locations (3):
- Taiwan (3):
  - Shuang Ho Hospital, New Taipei City
  - Taipei Medical University Hospital, Taipei
  - Wan Fang Hospital, Taipei

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] St Pierre K, Cashmore BA, Bolignano D, Zoccali C, Ruospo M, Craig JC, Strippoli GF, Mallett AJ, Green SC, Tunnicliffe DJ. Interventions for preventing the progression of autosomal dominant polycystic kidney disease. Cochrane Database Syst Rev. 2024 Oct 2;10(10):CD010294. doi: 10.1002/14651858.CD010294.pub3. PMID 39356039